CLINICAL TRIAL: NCT03947385
Title: A Phase 1/2 Study of IDE196 in Patients With Solid Tumors Harboring GNAQ/11 Mutations or PRKC Fusions
Brief Title: Study of IDE196 in Patients With Solid Tumors Harboring GNAQ/11 Mutations or PRKC Fusions
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: IDEAYA Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IDE196-001
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Uveal Melanoma; Cutaneous Melanoma; Colorectal Cancer; Other Solid Tumors
Keywords: Metastatic Uveal Melanoma; Uveal Melanoma; Protein Kinase C; Ophthalmology; Ocular Oncology; Darovasertib; IDE196; Ocular Melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma; Colorectal Neoplasms | interventions — Protein Kinase C; binimetinib; Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Dose Escalation Monotherapy (Enrollment Complete) (Experimental): IDE196 dosed orally, twice daily (BID) for each 28-day cycle
  Interventions: Drug: IDE196
- Dose Expansion Monotherapy (Enrollment Complete) (Experimental): RP2D in MUM and non-MUM tumors harboring GNAQ/11 mutations or PRKC fusions (cutaneous melanoma, CRC, other solid tumors)
  Interventions: Drug: IDE196
- Dose Escalation Binimetinib Combination (Enrollment Complete) (Experimental): IDE196 dosed orally, twice daily (BID) for each 28-day cycle and Binimetinib dosed orally, twice daily (BID) for each 28-day cycle
  Interventions: Drug: IDE196; Drug: Binimetinib
- Dose Expansion Binimetinib Combination (Enrollment Complete) (Experimental): RP2D in MUM and non-MUM tumors harboring GNAQ/11 mutations (cutaneous melanoma, CRC, other solid tumors)
  Interventions: Drug: IDE196; Drug: Binimetinib
- Dose Escalation Crizotinib Combination (Enrollment Complete) (Experimental): IDE196 dosed orally, twice daily (BID) for each 28-day cycle and Crizotinib dosed orally, twice daily (BID) for each 28-day cycle
  Interventions: Drug: IDE196; Drug: Crizotinib
- Dose Expansion Crizotinib Combination (Enrolling) (Experimental): MUM patients (previously treated or treatment naive) with human leukocyte antigen (HLA)-A*02:01 positive status.
  Includes a nested PK sub-study with Pravastatin (~22 participants) to evaluate the impact of pravastatin PK profiles after continuous dosing of IDE196.
  Includes a nested PK Cocktail DDI sub-study (~15 participants) to evaluate the impact on the PK of bupripion, repaglinide, flurbiprofen, omeprazole, midazolam, dabigatran etexilate, and the exposures of the OAT3 biomarker PDA by IDE196 in combination with crizotinib.
  Interventions: Drug: IDE196; Drug: Crizotinib
- Dose Optimization Crizotinib Combination (Enrollment Complete) (Experimental): IDE196 dosed orally, twice daily (BID) for each 28-day cycle and Crizotinib dosed orally, twice daily (BID) for each 28-day cycle
  Interventions: Drug: IDE196; Drug: Crizotinib
- Crizotinib Monotherapy with Crossover to Combination (Enrollment Complete) (Experimental): Crizotinib dosed orally, twice daily (BID) for each 28-day cycle until disease progression then IDE196 added and dosed orally, twice daily (BID) for each 28-day cycle
  Interventions: Drug: IDE196; Drug: Crizotinib

INTERVENTIONS:
Drug: IDE196 — IDE196 dosed orally, twice daily for each 28-day cycle
  Other Names: Protein Kinase C (PKC) Inhibitor
Drug: Binimetinib — Binimetinib dosed orally, twice daily for each 28-day cycle
  Other Names: MEKTOVI
  Arms: Dose Escalation Binimetinib Combination (Enrollment Complete); Dose Expansion Binimetinib Combination (Enrollment Complete)
Drug: Crizotinib — Crizotinib dosed orally, twice daily for each 28-day cycle
  Other Names: XALKORI
  Arms: Crizotinib Monotherapy with Crossover to Combination (Enrollment Complete); Dose Escalation Crizotinib Combination (Enrollment Complete); Dose Expansion Crizotinib Combination (Enrolling); Dose Optimization Crizotinib Combination (Enrollment Complete)

SUMMARY:
This is a Phase 1/2, multi-center, open-label basket study designed to evaluate the safety and anti-tumor activity of IDE196 in patients with solid tumors harboring GNAQ or GNA11 (GNAQ/11) mutations or PRKC fusions, including metastatic uveal melanoma (MUM), cutaneous melanoma, colorectal cancer, and other solid tumors.

Phase 1 (dose escalation - monotherapy) will assess safety, tolerability and pharmacokinetics of IDE196 via standard dose escalation scheme and determine the recommended Phase 2 dose. Safety and anti-tumor activity will be assessed in the Phase 2 (dose expansion) part of the study.

Phase 1 (dose escalation - binimetib combination) will assess safety, tolerability and pharmacokinetics of IDE196 and binimetinib via standard dose escalation scheme and determine the recommended Phase 2 dose. Safety and anti-tumor activity will be assessed in the Phase 2 (dose expansion) part of the study.

Phase 1 (dose escalation - crizotinib combination) will assess safety, tolerability and pharmacokinetics of IDE196 and crizotinib via standard dose escalation scheme and determine the recommended Phase 2 dose. Safety and anti-tumor activity will be assessed in the Phase 2 (dose expansion) part of the study. Evaluation of safety and efficacy across multiple doses may be explored in the dose optimization part of the study.

Crizotinib monotherapy with crossover to combination cohort may be assessed for safety and to show the contribution of each study drug to anti-tumor activity.

As of Protocol Amendment 10, Phase 1, Phase 2 dose expansion in IDE196 monotherapy, and Phase 2 dose expansion of IDE196 in combination with binimetinib have been fully enrolled. There were no patients enrolled in the crizotinib monotherapy cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥18 years of age and able to provide written informed consent
* Diagnosis of the following:

  o MUM: Uveal melanoma with histological or cytological confirmed metastatic disease. Metastatic disease may be treatment naïve or have progressed on or after most recent therapy. If the most recent therapy was an immune-oncology agent, PD must be confirmed.

  - If a patient is treatment naïve and human leukocyte antigen (HLA)-A*02:01 positive***, documentation is required to provide rationale why treatment with tebentafusp is not the ideal firstline treatment approach or of the patient's intolerance to tebentafusp.

  ***To be enrolled in the HLA-A*02:01 positive cohort, HLA status must be documented by test results from a CAP/CLIA-certified laboratory.
* Measurable disease per RECIST v1.1
* Eastern Cooperative Oncology Group ≤1 and expected life expectancy of > 3 months
* Adequate organ function at screening
* Adequate contraceptive measures for non-sterilized male and female patients of childbearing potential

Crizotinib Combination Additional Inclusion Criteria:

* Prior chemotherapy other therapies as applicable or major surgeries must have been completed at least 4 weeks prior to initiation of crizotinib
* Patients with preexisting peripheral neuropathy can be included if it is Grade 1 or lower, prior to initiation of crizotinib Biopsy-eligible patients
* Accessible lesion(s) that permit a total of at least two biopsies without unacceptable risk of a significant procedural complication.

Exclusion Criteria:

* Previous treatment with a PKC inhibitor
* Known MSI-H/dMMR tumors who have not previously received immune checkpoint inhibitors
* Known symptomatic brain metastases
* Adverse events from prior anti-cancer therapy that have not resolved
* Known acquired immunodeficiency syndrome (AIDS)-related illness, hepatitis B virus, or hepatitis C virus
* Active infection requiring ongoing therapy
* Recent surgery or radiotherapy
* Prior gastrectomy or upper bowel removal or any other gastrointestinal disorder or defect
* Females who are pregnant or breastfeeding
* Impaired cardiac function
* Treatment with prohibited medications that cannot be discontinued prior to study entry
* For patients receiving IDE196 powder-in-capsule (PIC) formulation or crizotinib, allergy to mammalian meat products and gelatin

Crizotinib Combination Additional Exclusion Criteria:

* Prior therapy directly targeting ALK, MET, or ROS1
* Spinal cord compression
* History of pneumonitis or interstitial lung disease
* History of syncope
* History of thromboembolic or cerebrovascular events ≤12 weeks prior to first dose of study treatment

PK Substudy (optional) with Pravastatin Additional Exclusion Criteria:

* Taken any dose of statin or inhibitor of organic anion transporting polypeptide within 7 days prior to enrollment in the study and cannot refrain from them through C2D1
* Taken drugs that interfere with the absorption, metabolism, or elimination of pravastatin
* Any contraindication associated to the use of statins or hypersensitivity component of pravastatin
* Active liver disease

DDI Cocktail Substudy Additional Exclusion Criteria:

* Treatment with bupropion, repaglinide, flurbiprofen, omeprazole, esomeprazole, midazolam, and dabigatran etexilate within 7 days prior to Cycle 1 Day -1.
* Intake of vitamin supplements containing Vitamin B6 (pyridoxine), grapefruit/grapefruit juice, or Seville orange juice within 7 days prior to Cycle 1 Day -1.
* Intake of any strong or moderate inhibitor of CYP2B6, CYP2CI, CYP2C9, CYP2C10 and OAT3 is prohibited within 7 days or within 5 half-lives, whichever is longer, of Cycle 1 Day -1.
* Moderate and strong inhibitors of CYP2A4/5 or P-gp are prohibited within 7 days, or within 5 half-lives, whichever is longer, of Cycle 1 Day -1.
* Intake of strong or moderate inducers of CYP3A4/5, CYP2B6, CYP2C9, CYP2C19, or OAT3 is prohibited during 15 days, or 5 half-lives, whichever is longer, prior to Cycle 1 Day -1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2019-06-28 (Actual); Primary Completion 2027-01-29 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity (DLT) | 28 days following first dose of IDE196 as monotherapy, in combination with Binimetinib, or in combination with Crizotinib
  Determine DLT of IDE196 as monotherapy, in combination with Binimetinib, or in combination with Crizotinib
Maximum Tolerated Dose (MTD) | 28 days following first dose of IDE196 as monotherapy, in combination with Binimetinib, or in combination with Crizotinib
  Determine MTD of IDE196 as monotherapy, in combination with Binimetinib, or in combination with Crizotinib
Recommended Phase 2 Dose (RP2D) as monotherapy, in combination with Binimetinib, or in combination with Crizotinib | Approx. 6 months
  Determine RP2D of IDE196 as monotherapy, in combination with Binimetinib, or in combination with Crizotinib
Incidence of Adverse Events | Approx. 8 months
  Safety and tolerability of IDE196 either as monotherapy, in combination with Binimetinib, or in combination with Crizotinib
Plasma Concentrations of IDE196 as monotherapy, in combination with Binimetinib, or in combination with Crizotinib | Approx. 6 months
  Pharmacokinetics of IDE196 as monotherapy, in combination with Binimetinib, or in combination with Crizotinib
Plasma Concentrations of Crizotinib administered in combination with IDE196 | Approx. 6 months
  Pharmacokinetics of Crizotinib in combination with IDE196
Plasma Concentrations of Binimetinib administered in combination with IDE196 | Approx. 6 months
  Pharmacokinetics of Binimetinib in combination with IDE196
Overall Response Rate (ORR) of IDE196 monotherapy, in combination with Binimetinib, and in combination with Crizotinib in Dose Expansion cohorts by Investigator response assessment | Approx. 8 months
  Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1) criteria
Duration of Response (DOR) of IDE196 monotherapy, in combination with Binimetinib, and in combination with Crizotinib in Dose Expansion cohorts by Investigator response assessment | Approx. 8 months
  RECIST v1.1
Phramacokinetic parameters of bupropion, hydroxybupropion, repaglinide, flurbiprofen, omeprazole, midazolam, total dabigatran, and the exposures of pyridoxic acid by IDE196 monotherapy and IDE196 in combination with Crizotinib | Approx. 8 months
  PK parameters of drug cocktail

SECONDARY OUTCOMES:
Progression Free Survival (PFS) of IDE196 monotherapy, in combination with Binimetinib, and in combination with Crizotinib in Dose Expansion cohorts by Investigator response assessment | Approx. 18 months
  RECIST v1.1
Overall Response Rate (ORR) of IDE196 monotherapy, in combination with Binimetinib, and in combination with Crizotinib in Dose Expansion cohorts and by prior treatment status (pretreated or treatment naive) by Investigator response assessment | Approx. 18 months
  Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1) criteria
Duration of Response (DOR) of IDE196 monotherapy, in combination with Binimetinib, and in combination with Crizotinib in Dose Expansion cohorts by prior treatment status (pretreated or treatment naive) by Investigator response assessment | Approx. 18 months
  RECIST v1.1
Disease Control Rate (DCR) by Investigator | Approx. 18 months
  RECIST v1.1

OTHER OUTCOMES:
Overall Survival | Approx. 18 months
  From date of First Dose to End of Follow-up
Anti-tumor activity (ORR/DOR/PFS) of IDE196 monotherapy, in combination with Binimetinib, and in combination with Crizotinib in Dose Expansion cohorts by Blinded Independent Review Committee (BICR) | Approx. 18 months
  RECIST v1.1
Anti-tumor activity (ORR/DOR/DCR) of IDE196 monotherapy, in combination with Binimetinib, and in combination with Crizotinib in phase 1 Dose Escalation cohorts by Investigator response assessment | Approx. 18 months
  RECIST v1.1
Anti-tumor activity (ORR/DOR/DCR) of IDE196 monotherapy, in combination with Binimetinib, and in combination with Crizotinib in pre-treated participants by Investigator response assessment | Approx. 18 months
  RECIST v1.1
Treatment-related gene signatures and/or molecular profiling | Approx. 18 months
  Modulation of gene signatures and/or molecular profiles
Treatment-related pharmacodynamic effect in all patients | Approx. 18 months
  Modulation of signaling proteins in PKC, MAPK, and MET pathways
Treatment-related changes in tumor tissue or cell-free DNA from blood | Approx. 18 months
  Modulation of tissue or cell-free DNA expression
Metabolite profile of IDE196 in plasma | Approx. 18 months
  Exploratory assessment of IDE196 metabolite profiling the plasma
Impact on pravastatin PK profile by IDE196 and Crizotinib combination | Approx. 18 months
  PK parameters of pravastatin

CONTACTS AND LOCATIONS:
Overall Officials: George Cole Jr., MD, Study Director — gcole@ideayabio.com
Locations (15):
- United States (12):
  - UCLA Medical Center, Los Angeles, California
  - San Francisco Oncology Associates, San Francisco, California
  - SCRI - Denver, Denver, Colorado
  - University of Iowa, Iowa City, Iowa
  - Cancer Hematology Centers Western Michigan, Grand Rapids, Michigan
  - Columbia University Medical Center - Herbert Irving Pavilion, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Cancer Center, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania
  - The Sarah Cannon Research Institute/Tennessee Oncology, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Westmead Hospital, Sydney, New South Wales
  - Queensland, Woolloongabba
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No